CLINICAL TRIAL: NCT00631228
Title: XIENCE V® Everolimus Eluting Coronary Stent System India Post-marketing Single-Arm Study
Acronym: XIENCE V India
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-378; REFCTRI000213, 21-10-2008 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; Angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: The group will be monitored to evaluate XIENCE V® EECSS continued safety and effectiveness during commercial use in real world settings.
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease
  Other Names: XIENCE V® Everolimus Eluting Coronary Stent System

SUMMARY:
XIENCE V® India is a prospective, open-label, multi-center, observational, single-arm study to evaluate XIENCE V® EECSS continued safety and effectiveness during commercial use in real world settings.

DETAILED DESCRIPTION:
Long term surveillance studies using a drug eluting stent (DES) may help elucidate mechanisms responsible for death, myocardial infarction, and late stent thrombosis risks not observed during controlled pre-market trials. This study will evaluate XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) performance in the "real world" when used by a broad group of physicians at a variety of health care facilities. Consequently, this protocol will include all consecutively enrolled patients in India who consent to participate and receive the XIENCE V® EECSS, which is expected to represent the range of clinical use during commercialization.

Adjunctive anti-platelet therapy is a critical factor in optimizing long term DES safety. Despite established guidelines that recommend 6-12 months dual antiplatelet therapy, patients with DES implants frequently stop taking their medication early. Consequently, XIENCE V® EECSS India Post-marketing Single-Arm Study (XIENCE V® India) follow-up will document patient adherence and persistence with adjunctive antiplatelet drug therapy at several time points throughout the study.

The long term safety and efficacy of the XIENCE V EECSS have been demonstrated in the SPIRIT FIRST trial up to 5 years, the SPIRIT II trial up to 4 years, and in the SPIRIT III Randomized Control Trial (RCT) up to 3 years. In addition, these pre-approval studies have shown low rates of Target Vessel Failure and Major Adverse Cardiac Events (MACE) that were observed to plateau or gradually decline after about 1 year and were consistently lower than the comparator arm of each study. This benefit in MACE is sustained for up to 5 years and is also independent of the first year results.

The post approval XIENCE V India study demonstrated that the use of the XIENCE EECSS in complex lesions in a real-world population resulted in 1 year MACE, Stent Thrombosis and Target Lesion Revascularization rates that are comparable to those of the previously mentioned pre-approval studies which included patients with more restricted inclusion / exclusion criteria.

Therefore, based on existing data from these trials, Abbott Vascular has decided to discontinue further follow up in the XIENCE V India study, from 5 years to after completion of the three year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient agrees to participate in this study by signing the EC approved informed consent form. Alternatively, the patient's legally authorized representative agrees to the patient's participation in this study and signs the informed consent form.

Exclusion Criteria:

* The inability to obtain an informed consent is an exclusion criterion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The group will be all consecutively enrolled patients in India treated by a broad group of physicians at a variety of health care facilities, who consent to participate and receive the XIENCE V® EECSS, which is expected to represent the range of clinical use during commercialization.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Stent thrombosis rates as defined by Academic Research Consortium (ARC) | Annually through to 3 years
Composite endpoint of cardiac death and myocardial infarction (MI) | at 1 year

SECONDARY OUTCOMES:
Composite rate of cardiac death and any MI (Q-wave and non Q-wave) | at 30, 180 days and at 2 and 3 years
Composite rate of all death and any MI (Q-wave and non Q-wave) | at 30, 180 days and at 2 and 3 years
Composite rate of cardiac death , any MI (Q-wave and non Q-wave) attributed to the target vessel, and target lesion revascularization (PCI and CABG) | at 30, 180 days and at 2 and 3 years
Death (cardiac death, vascular death, and non-cardiovascular death) | at 30, 180 days and at 2 and 3 years
Any MI (Q-wave and non Q-wave) | at 30, 180 days and at 2 and 3 years
Major bleeding complications | at 14, 30, 180 days and at 1, 2 and 3 years
Compliance and therapy interruptions with prescribed adjunctive antiplatelet therapy | at 14, 30, 180 days and at 1, 2 and 3 years
Revascularization (target lesion, target vessel [TVR], and non-target vessel) (PCI and CABG) | at 30, 180 days and at 1, 2 and 3 years
Clinical device and procedural success | Acute
Patient health status (symptoms, physical function, and quality of life) assessed by the Seattle Angina Questionnaire | at baseline, 180 days, and 1 year
Stent thrombosis | 24 hours (acute) and 30 days (sub-acute)
Composite rate of all death, any MI (Q-wave and non Q-wave) and any repeat revascularization (PCI and CABG) | 30, 180 days and 1, 2 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Seth, MD, Principal Investigator — Max Devki Devi Heart & Vascular Institute; Tejas Patel, MD, Principal Investigator — Krishna Heart Institute
Locations (17):
- India (17):
  - CARE Hospital, Hyderabaad, Andhra Pradesh
  - Krishna Heart Institute,, Hyderabad, Andhra Pradesh
  - Krishna Heart Institute, Ahmedabad, Gujarat
  - Jehangir Hospital, Pune, Pune
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Christian Medical Center (CMC), Vellore, Tamil Nadu
  - SAL Hospital And Medical Institute, Ahmedabad
  - Escorts Heart & Superspeciality Institute Ltd., Amritsar
  - Madras Medical Mission, Chennai
  - Apollo Hospital, Hyderabad
  - Heart & General Hospital, Jaipur
  - Lisie Heart Institute,Lisie Hosp., Kochi
  - Holy Family Hospital, Mumbai
  - Escorts Heart Institute & Research Centre, New Delhi
  - Fortis Hospital, New Delhi
  - Max Devki Devi Heart & Vascular Institute, New Delhi
  - Poona Hospital And Research Centre, Pune

REFERENCES:
- [Derived] Genereux P, Rutledge DR, Palmerini T, Caixeta A, Kedhi E, Hermiller JB, Wang J, Krucoff MW, Jones-McMeans J, Sudhir K, Simonton CA, Serruys PW, Stone GW. Stent Thrombosis and Dual Antiplatelet Therapy Interruption With Everolimus-Eluting Stents: Insights From the Xience V Coronary Stent System Trials. Circ Cardiovasc Interv. 2015 May;8(5):e001362. doi: 10.1161/CIRCINTERVENTIONS.114.001362. PMID 25940520